CLINICAL TRIAL: NCT01883089
Title: Ambivalence Model of Craving: Re-examining the Drinking-craving Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Robert Schlauch, Assistant Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Craving and Drinking
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Other (Other): Participants will be recruited to complete a 90 day daily monitoring study during which time will be invited to participate in a 4 week brief alcohol intervention during days 31-60 (i.e., second month).
  Interventions: Behavioral: Motivational Enhancement Therapy

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy

SUMMARY:
The current study combines both clinical trial and daily process methodology to examine the dynamic longitudinal relationships between daily approach and avoidance inclinations (i.e., craving) and drinking behaviors in those diagnosed with an Alcohol Use Disorder (AUD) prior to, during, and after receiving a brief alcohol intervention. It is hypothesized that daily avoidance inclinations will significantly moderate the effect of daily approach inclinations on drinking behaviors, and that significant increases in avoidance inclinations will be observed prior to treatment entry, followed by significant decreases in approach inclinations during treatment.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of alcohol dependence
* live within commuting distance of the program site,
* regular access to a phone to call into an IVR system and
* provide informed consent

Exclusion Criteria:

* acute psychosis or severe cognitive impairment
* current or previous treatment for an alcohol use disorder within the past 6 months,
* taking medications that may modify alcohol use,
* current drug use diagnosis other than nicotine or marijuana abuse,
* lack of sufficient familiarity with the English language to comprehend the recruitment and consent procedures, and
* legally mandated to attend treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Drinks per day | participants will be followed for the duration of the study, an expected average of 90 days
  Drinks consumed per day will be monitored daily over 90 days using interactive voice response systems (i.e., telephone call in).

SECONDARY OUTCOMES:
Approach inclinations | participants will be followed for the duration of the study, an expected average of 90 days
  Approach inclinations (desires to use alcohol) will be collected daily over 90 days using interactive voice response systems (i.e., telephone call in).
Avoidance inclinations | participants will be followed for the duration of the study, an expected average of 90 days
  Avoidance inclinations (desires to not use alcohol) will be collected daily over 90 days using interactive voice response systems (i.e., telephone call in).

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Schlauch, Phd, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Derived] Walsh BE, Dvorak RD, Ebbinghaus A, Gius BK, Levine JA, Cortina W, Schlauch RC. Disaggregating within- and between-person effects of affect on drinking behavior in a clinical sample with alcohol use disorder. J Psychopathol Clin Sci. 2023 Nov;132(8):1051-1059. doi: 10.1037/abn0000875. PMID 38010773